CLINICAL TRIAL: NCT05454384
Title: Evaluation of Consultation Contents Directed From a University Training and Research Hospital to an Oral and Maxillofacial Surgery Clinic
Brief Title: Consultation Contents of an Oral and Maxillofacial Surgery Clinic
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Aras Erdil, Asistant Professor Doctor, Tokat Gaziosmanpasa University
Other Study IDs: 21-KAEK-274
Record Dates: First submitted 2022-07-04; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Referral and Consultation
Keywords: Consultation, Dentistry; Forensic Odontology; Oncology; Oral and Maxillofacial Surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Forensic Medicine: The group of consultation records requested from the Department of Forensic Medicine
  Interventions: Other: Medical Record Examination
- Oncology: The group of consultation records requested from the Department of Oncology
  Interventions: Other: Medical Record Examination
- Neonatology: The group of consultation records requested from the Department of Neonatology
  Interventions: Other: Medical Record Examination
- Otorhinolaryngology: The group of consultation records requested from the Department of Otorhinolaryngology
  Interventions: Other: Medical Record Examination
- Neurology and Neurosurgery: The group of consultation records requested from the Department of Neurology and Neurosurgery
  Interventions: Other: Medical Record Examination
- Pediatrics: The group of consultation records requested from the Department of Pediatrics
  Interventions: Other: Medical Record Examination
- Emergency Medicine: The group of consultation records requested from the Department of Emergency Medicine
  Interventions: Other: Medical Record Examination
- Other Departments: The group of consultation records requested from the Departments such as Plastic and Reconstructive Surgery, Cardiovascular Surgery, Internal Medicine, Ophthalmology, Urology, Gastroenterology, Palliative Care, Pulmonology, Sleep Medicine, and Infectious Diseases.
  Interventions: Other: Medical Record Examination

INTERVENTIONS:
Other: Medical Record Examination — The patients' demographic features, related management and treatment process, the responses given to the consultations by OMFS clinic, the physicians' recommendations, the patient management, and the treatments applied by dentistry clinics were classified and recorded for statistical analyses.

SUMMARY:
This study aimed to evaluate conditions and indications in which a training and research hospital directs outpatient and inpatient consultations to an oral and maxillofacial surgery clinic and consider the expectations of physicians in the treatment and management of various conditions.

DETAILED DESCRIPTION:
The patients' consultation forms referred from the clinics and inpatient services of the Faculty of Medicine, Tokat Gaziosmanpasa University, between January 2013 and January 2022 were included in the current study via Enlil-Hospital Information Management System (Eskişehir, Turkey).

The consultation forms which were referred within the same institution or from the external institutions with written consultation notes and the patients with missing demographic data or consultation reports were excluded from the study.

The specific variables such as age, gender, the department in which consultations were requested, and for what purpose the patients were consulted were recorded and classified. During the patient management and treatment process, the responses given to the consultations by the Oral and Maxillofacial Surgery (OMFS) clinic, the physicians' recommendations, the patient management, and the treatments applied were classified and recorded for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* The patients' consultation forms were referred from the clinics and inpatient services of the Faculty of Medicine, Tokat Gaziosmanpasa University, to the Department of Oral and Maxillofacial Surgery of the same affiliation.

Exclusion Criteria:

* The consultation forms which were referred within the same institution or from the external institutions with written consultation notes and the patients with missing demographic data or consultation reports

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical records of patients who applied to Tokat Gaziosmanpasa University, Faculty of Medicine, Training and Research Hospital departments with the need for treatment were consulted with the Oral and Maxillofacial Surgery clinic of the same institution.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Reasons for Requesting Consultations | After completion of data collection, up to 3 weeks.
  The contents of the consultation requests were classified.
The Applied Treatments and Procedures | After completion of data collection, up to 3 weeks.
  The diagnosis and applied treatments and of the consulted patients in the department of oral and maxillofacial surgery clinic were analyzed.
Notable Consultation Requests | After completion of data collection, up to 3 weeks.
  The departments' consultation requests that frequently refer patients were analyzed regarding demographic variables, applied treatments, and examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Sefa Çolak, AssistProfDr, Study Director — Tokat Gaziosmanpasa University

IPD SHARING:
Plan to Share IPD: No
The data regarding participants were made available in the manuscript

REFERENCES:
- [Result] Sippli K, Rieger MA, Huettig F. GPs' and dentists' experiences and expectations of interprofessional collaboration: findings from a qualitative study in Germany. BMC Health Serv Res. 2017 Mar 7;17(1):179. doi: 10.1186/s12913-017-2116-4. PMID 28270205
- [Result] Avon SL. Forensic odontology: the roles and responsibilities of the dentist. J Can Dent Assoc. 2004 Jul-Aug;70(7):453-8. PMID 15245686